CLINICAL TRIAL: NCT00475475
Title: Sweetened Beverages and Food Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Mario Kratz, Research Assistant Professor, University of Washington
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 28740-A; 05-8515-A 03
Record Dates: First submitted 2007-05-16; First posted 2007-05-21 (Estimated); Last update posted 2012-05-02 (Estimated); Status verified 2012-04

CONDITIONS: Overweight; Obesity
Keywords: Overweight; Obesity; Appetite; Dietary sugars; Fructose; Glucose; Leptin; Insulin; Ghrelin
MeSH Terms: conditions — Overweight; Obesity; Insulin Resistance | interventions — Fructose; Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Fructose-sweetened beverage Subjects will be asked to drink 4 servings of a beverage sweetened with 100% fructose per day for 8 days, while consuming an ad libitum diet (same solid food for all three diet periods).
  Interventions: Behavioral: Fructose
- 2 (Experimental): Glucose-sweetened beverage Subjects will be asked to drink 4 servings of a beverage sweetened with 100% glucose per day for 8 days, while consuming an ad libitum diet (same solid food for all three diet periods).
  Interventions: Behavioral: glucose
- 3 (Placebo Comparator): Beverage sweetened with a non-caloric sweetener Subjects will be asked to drink 4 servings of a beverage sweetened with a non-caloric sweetener per day for 8 days, while consuming an ad libitum diet (same solid food for all three diet periods).
  Interventions: Behavioral: non-caloric sweetener

INTERVENTIONS:
Behavioral: Fructose — 25% of energy intake in the form of a fructose-sweetened beverage (arm 1), a glucose-sweetened beverage (arm 2), or an isovolumetric amount of a beverage sweetened with a non-caloric sweetener
  Arms: 1
Behavioral: glucose — 25% of energy intake in the form of a fructose-sweetened beverage (arm 1), a glucose-sweetened beverage (arm 2), or an isovolumetric amount of a beverage sweetened with a non-caloric sweetener
  Arms: 2
Behavioral: non-caloric sweetener — 25% of energy intake in the form of a fructose-sweetened beverage (arm 1), a glucose-sweetened beverage (arm 2), or an isovolumetric amount of a beverage sweetened with a non-caloric sweetener
  Arms: 3

SUMMARY:
The purpose of this study is to investigate whether beverages sweetened with fructose promote overconsumption of calories as compared to beverages sweetened with glucose or a non-caloric sweetener.

DETAILED DESCRIPTION:
The rise in the prevalence of obesity and type 2 diabetes mellitus has been linked to an increased consumption of sugar- and particularly fructose-sweetened beverages. Preliminary evidence suggests that this could be partly explained by the fact that the reduction in the intake of solid food is inadequate to compensate for additional energy taken up from these beverages. In addition, the type of sugar used to sweeten a beverage might have a considerable impact on the body's ability to adjust food intake properly. In particular, the consumption of fructose has been reported to reduce diurnal plasma glucose, insulin, and leptin concentrations, but increase diurnal ghrelin concentrations as compared to isocaloric amounts of glucose. As the plasma concentrations of glucose, insulin, leptin, and ghrelin are involved in the regulation of food intake and energy expenditure, this might impair the longer-term ability of the body to match food intake and energy expenditure to stabilize body weight.

To investigate whether the regular consumption of fructose-sweetened beverages leads to an increase in total energy intake, the investigators will enroll healthy normal-weight subjects into a controlled diet study using a double-blind randomized cross-over design. Each subject will complete three diet periods: solid food plus a beverage sweetened with fructose (A), solid food plus a beverage sweetened with glucose (B), solid food plus a beverage sweetened with a non-caloric sweetener (C). During each period, subjects will be provided with all their food for 8 days. These diets will consist of meals freshly prepared using regular food items typically found in the American diet. Solid food will be provided in excess of what the subjects are estimated to require. Subjects will be asked to eat as much of this food as they need to feel comfortably satiated, and to return all excess foods to the Nutrition Research Kitchen of the University of Washington (UW) General Clinical Research Center (GCRC). This returned food will be weighed to assess precisely the amount and type of food eaten by the subjects on each day of these diet periods. In addition to this solid food, subjects will be asked to drink a certain amount of a lemonade sweetened with either fructose (A), glucose (B), or a non-caloric sweetener (C). In groups A and B, the subjects will consume 25% of their estimated daily calorie requirement in the form of these sugar sweetened beverages, while the drink in period C will be of the same volume.

Subjects will be admitted to the GCRC on the morning of day 9 of each diet period for the measurement of resting metabolic rate by means of indirect calorimetry and blood draws for the measurement of fasting plasma concentrations of adipogenic hormones and plasma lipids. Furthermore, we will administer a standardized breakfast and draw blood before and 0, 15, 30, 60, 90, and 120 minutes after this meal to measure the postprandial plasma concentrations of insulin, ghrelin, and satiety signals. Following the last postprandial blood draw, we will serve another meal to measure ad libitum food intake. Our hypothesis is that subjects will have more appetite and consume more food after they have consumed the fructose-sweetened beverage for 8 days.

Primary outcome measures of this study will be the total energy consumed during the periods A, B, and C; the reduction in the intake of solid foods in periods A and B as compared to period C; and energy uptake during the ad libitum meal served on day 9 of each diet period. Secondary outcome measures will be resting energy expenditure and plasma concentrations of satiety and adiposity signals.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-25 years
* Body mass index: 20-25 kg/m2
* Weight stable to within 5 pounds for 6 months prior to entering the study
* Within 10 pounds of their lifetime maximum weight
* Ability to be admitted for 5 hours to the General Clinical Research Center of the University of Washington on three occasions
* Ability to provide informed written consent
* Willingness to consume only food provided by the Nutrition Research Kitchen of the University of Washington General Clinical Research Center for three periods of 8 days each

Exclusion Criteria:

* History of cardiovascular disease
* Presence of diabetes mellitus or impaired glucose tolerance (fasting glucose > 100 mg/dL)
* Presence of hypertension (blood pressure systolic/diastolic higher than 140/90)
* Presence of phenylketonuria
* Presence of fructose malabsorption or hereditary fructose intolerance
* Presence of another chronic or psychiatric illness
* Use of anabolic steroids, glucocorticoids, warfarin, beta-blockers, antidepressants, or lipid-lowering agents
* Use of antibiotic drugs within 3 months of enrollment into the study
* Use of tobacco products
* Pregnancy or female subject not using contraception
* Regular intense exercise (> 3 hour per week)
* Vegetarian or extreme dietary preferences
* Alcohol consumption of more than 2 drinks per day
* Presence of eating disorder
* History of frequent attempts at weight loss
* Currently dieting or in a weight control program
* Recent blood donation or enrolled in other research which requires blood sampling
* Presence or history of anemia

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2007-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Total energy consumed in the three diet periods. | 8 days in each period

SECONDARY OUTCOMES:
Resting energy expenditure | After 8 days of each dietary phase
  Resting energy expenditure, as measured by indirect calorimetry.
Fasting and postprandial plasma concentrations of satiety and adiposity signals. | After 8 days of each dietary phase
  We will measure the fasting plasma concentration of leptin, adiponectin, ghrelin, insulin, glucagon-like peptide 1 (GLP-1), peptide YY (PYY), cholecystokinin (CCK), amylin, and oxyntomodulin, and the change in these endpoints in the two ours after a standardized meal has been consumed.
Fasting and postprandial plasma lipid and lipoprotein concentrations. | After 8 days of each dietary phase
  We will measure the fasting plasma concentrations of total cholesterol, LDL-cholesterol, HDL-cholesterol, triglycerides, and free fatty acids, as well as the changes in these endpoints in the two hours following a standardized meal. We will also measure the fatty acid composition in the plasma phospholipids, and the free fatty acid fraction of plasma.
Fasting plasma concentrations of inflammatory mediators. | After 8 days of each dietary phase
  We will measure the fasting plasma concentrations of C-reactive protein (high sensitivity assay), interleukin-6 (IL-6), and the soluble tumor necrosis factor alpha receptors I & II.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Kratz, Ph.D., Principal Investigator — University of Washington
Locations (1):
- University of Washington General Clinical Research Center, Seattle, Washington, United States

REFERENCES:
- [Derived] Kuzma JN, Cromer G, Hagman DK, Breymeyer KL, Roth CL, Foster-Schubert KE, Holte SE, Callahan HS, Weigle DS, Kratz M. No difference in ad libitum energy intake in healthy men and women consuming beverages sweetened with fructose, glucose, or high-fructose corn syrup: a randomized trial. Am J Clin Nutr. 2015 Dec;102(6):1373-80. doi: 10.3945/ajcn.115.116368. Epub 2015 Nov 4. PMID 26537945